CLINICAL TRIAL: NCT01054092
Title: Long-term Study of ASP1941 - A Phase III, Open-Label, Uncontrolled, Monotherapy Study to Assess the Long-term Safety, Tolerability and Efficacy of ASP1941 in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess the Long-term Safety and Efficacy of ASP1941 in Japanese Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1941-CL-0121
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Blood glucose; ASP1941; Food effect; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- before meal group (Experimental): ASP1941 will be administered before meal
  Interventions: Drug: ipragliflozin
- after meal group (Experimental): ASP1941 will be administered after meal
  Interventions: Drug: ipragliflozin

INTERVENTIONS:
Drug: ipragliflozin — oral
  Other Names: ASP1941

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of ASP1941 in patients with type 2 diabetes mellitus. The second objectives are to compare the efficacy and pharmacokinetics of ASP1941 administered before or after food intake.

DETAILED DESCRIPTION:
Subject will be randomized into either ASP1941 before meal or ASP1941 after meal groups. Subjects will undergo a screening period before entering the long-term treatment. Dosage may be increased during the treatment period if subjects fulfill increasing criteria and the investigators adjudicate that no impact for subjects safety.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients for at least 12 weeks
* HbA1c value between 6.5 and 9.5%
* Body Mass Index ( BMI )20.0 - 45.0kg/m2

Exclusion Criteria:

* Type 1 diabetes mellitus patients
* Serum creatinine > upper limit of normal
* Proteinuria (albumin/creatinine ratio > 300mg/g)
* Dysuria and/or urinary tract infection, genital infection
* Significant renal, hepatic or cardiovascular diseases
* Severe gastrointestinal diseases
* Proliferative diabetic retinopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-01-14 (Actual); Primary Completion 2011-07-22 (Actual); Study Completion 2011-07-22 (Actual)

PRIMARY OUTCOMES:
HbA1c | For 52 weeks

SECONDARY OUTCOMES:
Fasting plasma glucose | For 52 weeks
Fasting serum insulin | For 52 weeks
Plasma levels of ASP1941 for population PK analysis | For 52 weeks
Safety assessed by adverse events, vital signs laboratory tests and 12-lead ECGs | For 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Tōhoku

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=106